CLINICAL TRIAL: NCT00413647
Title: A Phase I Study to Evaluate the Safety, Biodistribution and Radiation Dosimetry of CardioPET™ as a PET Tracer for Detection of Coronary Artery Disease
Brief Title: A Phase I Study in Healthy Volunteers to Evaluate the Safety of CardioPET™ in Detection of Coronary Artery Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fluoropharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CardioPET P-01
Record Dates: First submitted 2006-12-18; First posted 2006-12-20 (Estimated); Last update posted 2013-06-12 (Estimated); Status verified 2013-06

CONDITIONS: Coronary Artery Disease
Keywords: CardioPET; Coronary Artery Disease; Electrocardiogram; Radiation Dosimetry
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CardioPET (Experimental)
  Interventions: Drug: CardioPET

INTERVENTIONS:
Drug: CardioPET

SUMMARY:
Safety and dosimetry of CardioPET™ will be evaluated in normal healthy volunteers and CAD subjects both male and female between the ages of 50-85. Nine normal controls will undergo repeated whole body imaging for biodistribution and dosimetry estimation. Six other normal healthy subjects will undergo heart imaging only. Six CAD subjects will undergo heart imaging only.

DETAILED DESCRIPTION:
CardioPET™ is a modified fatty acid (MFA) that closely resembles naturally-occurring free fatty acids (FFAs) in the human body.

Study Procedures:

Visit 1: Screening - Eligibility determination

Visit 2: Injection and PET Imaging

Visit 3: Follow-up Visit

ELIGIBILITY:
Inclusion Criteria:

Normal Healthy Volunteers:

* Subject must provide written informed consent prior to any study related procedures
* Subjects must be between the ages of 50 and 85 years of age.

Coronary Artery Disease (CAD) subjects:

* Subjects must provide written informed consent prior to any study related procedures;
* Subjects must be ≥ 50 and ≤ 85 years of age;
* Subject must have history of CAD documented by an exercise stress Myocardial Perfusion Imaging (MPI) study within 6 months documenting myocardial infarct without ischemia.

Exclusion Criteria:

Normal Healthy Volunteers:

* Any clinically significant acute or unstable physical or psychological disease based on medical history or screening physical examination
* Any clinically significant abnormality in the screening laboratory tests or ECG
* Fasting blood glucose level over 120 mg/dl
* Any exposure to any investigational drugs with four(4)weeks prior to Visit 1
* Any exposure to radiopharmaceuticals within four(4)weeks prior to the date of Visit 1
* Any new prescription medications within four(4)weeks of Visit 1
* Subject has a Positive(+)Serum and/or Urine Pregnancy Test or is lactating, or the possibility of pregnancy cannot be ruled out prior to dosing. There are standard pregnancy procedures for use of radiopharmaceuticals in research at MGH

Coronary Artery Disease (CAD) Subjects:

* Subject has a Positive (+) Serum and/or Urine Pregnancy Test or is lactating, or the possibility of pregnancy cannot be ruled out prior to dosing;
* Any clinically significant acute or unstable physical or psychological disease judged by the investigators based on medical history or screening physical examination;
* Coronary artery bypass graft (CABG) within 1 year;
* Percutaneous coronary intervention (PCI), with stent placement within three months;
* Blood pressure over 180/100;
* Acute changes in ECG;
* Cardiac ischemia identified by MPI stress test;
* Recent (within 3 months) cardiac arrest, unstable angina, myocardial infarction, cerebro-vascular accident (CVA), any general anesthesia procedure, any surgical procedures;
* Any implanted pacemaker or defibrillator use within the last three months;
* Inability to remain in camera for approximately 60 minutes (Smokers and COPD are included as long as they can breath in PET camera and not taking O2 through nasal canola);
* History of Diabetes Mellitus;
* Serum creatinine > 2 mg/dL;
* All cancer and or chemotherapy patients;
* Body Mass Index (BMI) is over 35;
* Any exposure to any investigational drugs or medical device within four (4) weeks prior to imaging study;
* Any exposure to radiopharmaceuticals within four (4) weeks prior to the date of imaging study;
* High daily alcohol consumption over 4 alcohol drinks per day.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2006-09; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Change in vital signs. Change in physical examination. Change in ECG. Change in 24-hour Holter. Change in dosimetry (blood and urine)measured at time 0 (immediately folloing injection), 1, 5, 15, 30, 60, and 90 minutes. Adverse event assessment. | Screening, Pre-dose, Baseline, Day 1, Pre-, Post-Dose 0, 24-48 hours and 7 days (Adverse events).
  Normal healthy volunteers for whole body imaging group and NHV and Coronary Artery Disease (CAD)undergoing cardiac imaging.

SECONDARY OUTCOMES:
Performance characteristics of CardioPET as a PET tracer for myocardial imaging. | 0, 1 min, 5 min, 15 min, 30 min, 60 min, and 90 min.
  Normal healthy volunteers and CAD subjects for Cardiac Imaging Only.
Evaluation and optimization of the methods of image acquisition, output processing, display, reconstruction, and imaging data | Baseline, 15 second time frames for first 2 minutes, 1 min. time frame for next 8 min., 2 min frames for remainder of 60 min study.

CONTACTS AND LOCATIONS:
Overall Officials: Alan J. Fischman, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States